CLINICAL TRIAL: NCT00544310
Title: A Prospective, Controlled, Randomized, Multi-Center, Exploratory Pilot Study Evaluating the Safety and Potential Trends in Efficacy of Adhexil
Brief Title: Pilot Study Evaluating the Safety and Potential Trends in Efficacy of Adhexil
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OMRIX Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: AA-GYN-001
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Bilateral Ovarian Disease

ARMS (1):
- 1 (Experimental): Post surgery adhesion prevention treatment
  Interventions: Biological: Anti adhesion agent

INTERVENTIONS:
Biological: Anti adhesion agent — Adhesions prevention
  Other Names: Adhexil

SUMMARY:
The objective is to evaluate the safety and initial efficacy of the Omrix Anti-Adhesion (AA) kit, Adhexil™ in preventing and/or reducing post-operative adhesions in patients undergoing surgery involving the ovaries.

DETAILED DESCRIPTION:
Adhexil™ contains the components that form the anti-adhesive barrier, BAC and Thrombin. Thrombin is a sterile solution, containing highly purified human thrombin. BAC is a sterile, solution whose principal component is a concentrate of human fibrinogen. Adhexil™ is supplied in two vials and an application device.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-45 years at screening
* Patients undergoing elective laparoscopic surgery due to known or suspected bilateral ovarian disease

Exclusion Criteria:

* Pregnant (including ectopic pregnancy) or breastfeeding patient
* Patients with a documented diagnosis of cancer
* Patients with a lymphatic, hematologic or coagulation disorder
* Patients with a known or suspected hypersensitivity to blood, blood products or any constituent of Adhexil™
* Patients who are immunocompromised, possess autoimmune disorders, or who are routinely taking anticoagulants.
* Patients who have participated in another clinical study within 30 days of enrolment.
* Investigator's opinion that the patient is medically unfit or would be at major risk if enrolled into the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25
Dates: Start 2008-01; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Preventing and/or reducing post-operative adhesions in patients undergoing surgery involving the ovaries

CONTACTS AND LOCATIONS:
Locations (4):
- New York, New York, United States
- Duisburg, Germany
- Valencia, Spain
- Oxford, United Kingdom